CLINICAL TRIAL: NCT04619173
Title: Additional Effects of Thoracic Manipulation in Patients With Adhesive Capsulitis.
Brief Title: Additional Effects of Thoracic Manipulation in Adhesive Capsulitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00675 Ubaidullah Bilal
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Frozen Shoulder
Keywords: Frozen Shoulder; Thoracic Manipulation
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic manipulation (Experimental): additional thoracic manipulation along with hotpack, transcutaneous electrical nerve stimulation ,serratus anterior,pectoralis major,minor, posterior capsular stretches..
  Interventions: Other: Thoracic manipulation
- Conventional Physical Therapy Program (Active Comparator): hot pack transcutaneous electrical nerve stimulation, serratus,anterior,pectoralis major, minor, posterior capsular stretches.
  Interventions: Other: Conventional physical therapy Program

INTERVENTIONS:
Other: Thoracic manipulation — hot pack ,transcutaneous electrical nerve stimulation and manipulation along with stretching'
  Arms: Thoracic manipulation
Other: Conventional physical therapy Program — hot pack ,transcutaneous electrical nerve stimulation and stretching
  Arms: Conventional Physical Therapy Program

SUMMARY:
The aim of this study is to measure the additional effects of thoracic manipulation on pain and restricted shoulder mobility and reducing disability in patients with adhesive capsulitis. A randomized control trail is conducting at Helping hand institute of rehabilitation sciences Mansehra. Patients diagnosed with frozen shoulder were randomized into 2 groups i.e. Group A (n=16) and Group B(n=16) with the help of lottery method. Group A would receive conventional therapy including hot pack, transcutaneous electrical nerve stimulation, stretches and facilitation techniques Group B would receive thoracic manipulation along with hot pack and TENS, stretches and facilitation techniques. The total treatment time is 2 weeks with three sessions per week making a total of 6 sessions.

Baseline assessment on 1st visit. 2nd assessment on 6th visit. 3rd assessment on follow up after 3 weeks would be done. The study duration is 6 months. Purposive non probability sampling technique applied. Only 40 to 60 years participants with adhesive capsulitis are including in this trial. Tools use in this study are visual analogue scale (VAS), bubble inclinometer and (disability of arm, shoulder and hand) questionnaire. Data analyzed through statistical package of social sciences version 25.

DETAILED DESCRIPTION:
Frozen shoulder is a widespread disabling condition which causes significant disability. In spite of hundred years of treating this condition the clarity, diagnosis, pathology and most effectual treatments are still need to be explored.It is characterized by the impulsive onset of pain, inflexibility and restricted range of motion at the shoulder joint. The pathophysiology of frozen shoulder is not exactly known. However it is generally supposed that a combination of contracture of capsule, rotator cuff tendon fibrosis, sub-scapular depression and the coraco-humeral ligament lead to comprehensive movement restriction at the glenohumeral joint. Frozen shoulder is considered to have an occurrence of 3%-5% in the common population and up to 20% in those with diabetes mellitus. Between the ages of 40 and 60 it is most prevalent and is almost not found in ages below that and in persons who work manually. It is somewhat more common in women then man. Bilateral frozen shoulder occurs in 14% of population and up to 20% of population will develop some degree of related symptoms in the other shoulder. the most common associated risk factor for developing the frozen shoulder is diabetes mellitus, and a patient with diabetes has 10%-20% risk of developing frozen shoulder.

Thoracic spine manipulation has received growing attention in treating the patients with shoulder pain. Recent studies have shown that thoracic manipulation is an effective combination therapy for patients with shoulder pain. The position of thoracic spine significantly have an effect on shoulder joint and shoulder kinematics during movement on different planes as there is decreased muscle force when a person is in a slouch position. Thoracic Spine manipulation is a treatment choice by the number of health professionals especially the physical therapist. Literature defines thoracic manipulation as highly practiced and skilled passive thrust to joints and adjacent structures and soft tissues at variable intensity consisting of small amplitude and high velocity therapeutic movements at thoracic spine including cervicothoracic junction. Much of the recent studies are focusing on the relationship of thoracic spine to other body regions such as neck and shoulder rather than thoracic spine itself this phenomenon is described as regional interdependence.although cervical spine manipulation has also improve pain and disability in patients with non-specific shoulder pain but have some evidence of thrust complications relating to cervical spine. Similar neurophysiologic associations are documented with thoracic spine manipulation in relation with shoulder pain with less complications and thrust risk.

Spinal manipulation of the thoracic spine can be an effective intervention for treating patients with shoulder pain or dysfunctions. Treatment protocols focusing the thoracic spine must be added to the intervention of rehabilitation of patients with shoulder pain in clinical practice. In common clinical practice a series of thoracic hypomobility has been noticed at the T1-T3 spinal segments or the T3-T5 segments in patients with shoulder pathologies. In literature manipulation of thoracic regions has been shown to produce improvement in upper extremity blood flow and circulation. Researches related to thoracic spine manipulation is signifying a association between manipulation of the thoracic spine and enhancement in shoulder function and potency. Thus the purpose of the study is to evaluate the possible effect of thoracic manipulation on shoulder range of motion and function in combination with conventional intervention for the individuals with frozen shoulder.

Thoracic spine thrust manipulation provided a statistically significant decrease in self-reported pain measures and disability in patients with Shoulder impingement syndrome. Thoracic spine and upper rib manipulative therapy is associated with improvement in shoulder pain and ROM immediately following intervention in patients with a primary complaint of shoulder pain. Thoracic spine manual therapy accelerated recovery and reduced pain and disability in patients having nonspecific shoulder pain (NSSP). Thoracic and rib manipulation is effective in relieving pain and improving range of motions and reducing disability in frozen shoulder patients. Cervical thoracic junction and upper thoracic spine manipulations in combination with traditional physical therapy will decrease pain, increase range of motion, and increase function in patients suffering from internal impingement syndrome more than patients who received traditional physical therapy treatment and posterior and inferior mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Adhesive capsulitis (Stage II and III)
* Bilateral or unilateral involvement
* Thoracic spine hypomobility

Exclusion Criteria:

* Any previous Surgery on the affected shoulder.
* Recent trauma to shoulder complex.
* Thoracic outlet syndrome.
* Cervical symptoms (tingling, numbness).
* Rotator cuff tears of affected shoulder.
* Fractures involving shoulder complex.
* Osteoporosis of spine.
* Ankylosing spondylitis

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS): | 3 weeks
  Visual analogue scale is a simple and frequently used method for the assessment of variations in intensity of pain. The VAS consists of a 10cm horizontal line with the words "no pain" and "worst pain" at the line's end. VAS is a reliable and valid tool to reliable and valid tool to measure pain intensity measure pain intensity. Changes from the baseline will be measured and at 4th week and then at 6th week
Bubble Inclinometer | 3 weeks
  Bubble Inclinometer is used to measure range-of-motion (ROM).
(Disabilities of the Arm, Shoulder and Hand) questionnaire: | 3 weeks
  The Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure is a 30-item, self-report questionnaire that measures physical function and symptoms in people with musculoskeletal disorders of the upper limb.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Helping Hand Institute of Rehabilitation Sciences, Mānsehra, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uppal HS, Evans JP, Smith C. Frozen shoulder: A systematic review of therapeutic options. World J Orthop. 2015 Mar 18;6(2):263-8. doi: 10.5312/wjo.v6.i2.263. eCollection 2015 Mar 18. PMID 25793166
- [Background] Riley SP, Bialosky J, Cote MP, Swanson BT, Tafuto V, Sizer PS, Brismee JM. Thoracic spinal manipulation for musculoskeletal shoulder pain: Can an instructional set change patient expectation and outcome? Man Ther. 2015 Jun;20(3):469-74. doi: 10.1016/j.math.2014.11.011. Epub 2014 Dec 2. PMID 25543999
- [Background] Kebaetse M, McClure P, Pratt NA. Thoracic position effect on shoulder range of motion, strength, and three-dimensional scapular kinematics. Arch Phys Med Rehabil. 1999 Aug;80(8):945-50. doi: 10.1016/s0003-9993(99)90088-6. PMID 10453773
- [Background] Walser RF, Meserve BB, Boucher TR. The effectiveness of thoracic spine manipulation for the management of musculoskeletal conditions: a systematic review and meta-analysis of randomized clinical trials. J Man Manip Ther. 2009;17(4):237-46. doi: 10.1179/106698109791352085. PMID 20140155
- [Background] Peek AL, Miller C, Heneghan NR. Thoracic manual therapy in the management of non-specific shoulder pain: a systematic review. J Man Manip Ther. 2015 Sep;23(4):176-87. doi: 10.1179/2042618615Y.0000000003. PMID 26917935
- [Background] Boyles RE, Ritland BM, Miracle BM, Barclay DM, Faul MS, Moore JH, Koppenhaver SL, Wainner RS. The short-term effects of thoracic spine thrust manipulation on patients with shoulder impingement syndrome. Man Ther. 2009 Aug;14(4):375-80. doi: 10.1016/j.math.2008.05.005. Epub 2008 Aug 15. PMID 18703377
- [Background] Alptekin HK, Aydin T, Iflazoglu ES, Alkan M. Evaluating the effectiveness of frozen shoulder treatment on the right and left sides. J Phys Ther Sci. 2016 Jan;28(1):207-12. doi: 10.1589/jpts.28.207. Epub 2016 Jan 30. PMID 26957759
- [Background] Kraal T, The B, Boer R, van den Borne MP, Koenraadt K, Goossens P, Eygendaal D. Manipulation under anesthesia versus physiotherapy treatment in stage two of a frozen shoulder: a study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2017 Oct 11;18(1):412. doi: 10.1186/s12891-017-1763-2. PMID 29020962
- [Background] Eljabu W, Klinger HM, von Knoch M. Prognostic factors and therapeutic options for treatment of frozen shoulder: a systematic review. Arch Orthop Trauma Surg. 2016 Jan;136(1):1-7. doi: 10.1007/s00402-015-2341-4. Epub 2015 Oct 17. PMID 26476720
- [Background] Wu WT, Chang KV, Han DS, Chang CH, Yang FS, Lin CP. Effectiveness of Glenohumeral Joint Dilatation for Treatment of Frozen Shoulder: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Sci Rep. 2017 Sep 5;7(1):10507. doi: 10.1038/s41598-017-10895-w. PMID 28874727
- [Background] Cao DZ, Wang CL, Qing Z, Liu LD. Effectiveness of extracorporeal shock-wave therapy for frozen shoulder: A protocol for a systematic review of randomized controlled trial. Medicine (Baltimore). 2019 Feb;98(7):e14506. doi: 10.1097/MD.0000000000014506. PMID 30762780
- [Background] McClure P, Balaicuis J, Heiland D, Broersma ME, Thorndike CK, Wood A. A randomized controlled comparison of stretching procedures for posterior shoulder tightness. J Orthop Sports Phys Ther. 2007 Mar;37(3):108-14. doi: 10.2519/jospt.2007.2337. PMID 17416125
- [Background] Strunce JB, Walker MJ, Boyles RE, Young BA. The immediate effects of thoracic spine and rib manipulation on subjects with primary complaints of shoulder pain. J Man Manip Ther. 2009;17(4):230-6. doi: 10.1179/106698109791352102. PMID 20140154
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Schilling DT, Mallace AJ, Elazzazi AM. SHOULDER RANGE OF MOTION CHARACTERISTICS IN DIVISION III COLLEGIATE SOFTBALL AND BASEBALL PLAYERS. Int J Sports Phys Ther. 2019 Sep;14(5):770-784. PMID 31598415
- [Background] Hammond A, Prior Y, Tyson S. Linguistic validation, validity and reliability of the British English versions of the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire and QuickDASH in people with rheumatoid arthritis. BMC Musculoskelet Disord. 2018 Apr 16;19(1):118. doi: 10.1186/s12891-018-2032-8. PMID 29661183